CLINICAL TRIAL: NCT06308809
Title: Effect of PNF Training as an Intervention for Functional Ankle Instability in College Student
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ma Shuzhen (Other)
Responsible Party: Sponsor-Investigator, Ma Shuzhen, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Shuzhen Ma
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Behavior
Keywords: adolescent population; PNF training
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
  - Page 2 of 5 [DRAFT] -In order to avoid mutual interference between the experimental group and the control group, a blinding method needs to be used in the study. In this study, a single blind experiment will be conducted to blind the participating athletes.
  During the sample grouping process, participating athletes will not know the specific grouping situation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF training group (Experimental): The experimental group will undergo 60 minutes of PNF training.
  Interventions: Other: PNF training
- Control training group (Other): The control group will follow the curriculum standards set by the Sports University.
  Interventions: Other: PNF training

INTERVENTIONS:
Other: PNF training — The subjects underwent rehabilitation training for 8 weeks, three times a week (Monday, Wednesday and Friday, 6:00 PM to 10:00 PM in the Physical Education College of Guangxi Normal University), and the rehabilitation training time was about 40-45 minutes per person. Before each rehabilitation training, the subjects warmed up the ankle and lower leg muscles for 5 minutes, followed by the corresponding rehabilitation training for 30-35 minutes, and relaxed the ankle and lower leg muscles for 5 minutes after the training.

SUMMARY:
The lower limb stability test was carried out by MicroSwing 6.0 gravity center moving trajectory tester made in Germany.

DETAILED DESCRIPTION:
The test steps and methods are as follows:

1. Before the test, arrange the subjects to be familiar with the lower limb stability test system and test environment, and master the test method.
2. The subject stands barefoot and one foot in the center of the center of gravity movement trajectory tester, with his hands placed on his sides naturally, and maintains his body balance for 30 seconds.
3. Record data of the test system.
4. The measurement was repeated three times with a time interval of 5min. Collect the test data of the center of gravity moving trajectory tester, including swing frequency, coordination coefficient and stability coefficient, and get the best results of the three tests. The smaller the oscillation frequency and coordination coefficient are within a certain range, the better the stability is. The greater the value of stability coefficient is within a certain range, the better the stability is.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral functional ankle instability;
2. Have not received formal rehabilitation treatment or informal rehabilitation treatment within the past month;
3. Voluntarily accept the treatment in this study and ensure to complete the training tasks arranged by the therapist;
4. Aged between 18 and 23 years old;

Exclusion Criteria:

1. Does not meet the above diagnostic criteria;
2. Ankle pain caused by infectious diseases;
3. suffering from severe neurological diseases;
4. Soft tissue damage near the ankle joint;
5. Other joints outside the ankle are unstable.

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
CAIT score | Baseline, post-test after 8 weeks
  CAIT consists of 9 questions with a total of 30 points, scoring ≦27 points for diagnosis of functional ankle instability, 28 points and above for diagnosis of non-functional ankle instability.
  1. Before issuing the questionnaire, explain the contents of the questionnaire to the subjects in detail, and the subjects fill in the questionnaire truthfully according to their own situation.
  2. The CAIT score of the subjects was calculated and recorded.
  3. If you fill in the questionnaire incorrectly, you need to fill it again and keep a record
Lower limb stability test | Baseline, post-test after 8 weeks
  The lower limb stability test was carried out by MicroSwing 6.0 gravity center moving trajectory tester made in Germany. The test steps and methods are as follows:
  1. Before the test, arrange the subjects to be familiar with the lower limb stability test system and test environment, and master the test method.
  2. The subject stands barefoot and one foot in the center of the center of gravity movement trajectory tester, with his hands placed on his sides naturally, and maintains his body balance for 30 seconds.
  3. Record data of the test system.
  4. The measurement was repeated three times with a time interval of 5min. Collect the test data of the center of gravity moving trajectory tester, including swing frequency, coordination coefficient and stability coefficient, and get the best results of the three tests.
Star offset balance test | Baseline, post-test after 8 weeks
  The subjects stood in the center of the star chart with the affected side foot as the supporting foot, with bare feet and one foot in the center. The healthy side foot was extended forward, outward front, outer front, outer back, back, inner back, inner and inner front respectively to the farthest distance as far as possible. The supporting foot was extended in the counterclockwise direction when the left foot was used, and the supporting foot was extended in the clockwise direction when the right foot was used. The subject withdrew the non-supporting foot and resumed standing with both feet and rested for 5 seconds. The data of each extension of the subject was recorded, and the farthest score was measured three times. The furthest results in each direction were standardized with the subjects' lower limb length, and the data were recorded.
  (4) The furthest scores in each direction were standardized with the subjects' lower limb length, and the data were recorded.
Muscle strength test | Baseline, post-test after 8 weeks
  MicroFET2 hand-held muscle strength tester made in Germany was used for muscle strength test. The test steps and methods are as follows:
  1. Before the test, arrange the subjects to be familiar with the handheld muscle strength test system and test environment, and master the test method.
  2. The subject took off his shoes and socks and lay on his back on the recovery bed with his hands naturally placed on his chest. The muscle strength of the subject's dorsalis, plantar flexus, varus and valgus were tested respectively.
  3. Record data of the test system.
  4. The measurement was repeated 5 times in each direction of movement. The test data of handheld muscle strength tester were collected, including the muscle strength of ankle dorsiflexion, plantar flexion, varus and valgus, and the best results of 5 tests were obtained.

IPD SHARING:
Plan to Share IPD: No